CLINICAL TRIAL: NCT01513837
Title: PREVALENCIA, GRAVEDAD E IMPACTO DE LA RINITIS Y DE LA SINUSITIS SEGÚN EL NIVEL DE GRAVEDAD Y CONTROL DEL ASMA (PROYECTO IRIS-ASMA)
Brief Title: Rinitis y Sinusitis según la Gravedad Del Asma
Acronym: IRIS-ASMA
Status: Completed | Type: Observational
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Sociedad Española de Neumología y Cirugía Torácica (Other)
Responsible Party: Principal Investigator, José Antonio Castillo Vizuete, MD, Sociedad Española de Neumología y Cirugía Torácica
Other Study IDs: SEPARALAT-1010-PII
Record Dates: First submitted 2012-01-17; First posted 2012-01-20 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

SUMMARY:
Based on the evidence for the "common pathway" in asthma presentation, our working hypothesis is that asthma severity and lack of control are related to the prevalence and severity of nasal and sinusal inflammatory pathology, and especially to chronic rhinosinusitis with nasal polyps.

DETAILED DESCRIPTION:
Primary objective: To assess the prevalence and severity of rhinitis and rhinosinusitis, with or without nasal polyposis, in asthmatic patients depending on severity of their disease.

Secondary objectives:

To assess the impact of nasal and sinusal pathology on asthma control.

To correlate asthma severity to rhinitis and rhinosinusitis.

To compare the potential association between chronic rhinosinusitis, with and without nasal polyposis, and asthma severity, and to detect radiographic differences, markers of atopy, and pulmonary function.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes aged 18-70 years attending outpatient clinics diagnosed with asthma at least one year before. GINA/GEMA criteria will be used to diagnose asthma and to rate its severity.

Exclusion Criteria:

* Illiterate patients;
* very severe, disabling comorbidity;
* prior non-inflammatory nasosinusal disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitals in Spain and Latin America
Sampling Method: Probability Sample
Enrollment: 450 (Estimated)
Dates: Start 2011-03; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Sociedad Española de Neumología y Cirugía Torácica (SEPAR), Barcelona, Catalonia, Spain